CLINICAL TRIAL: NCT06184243
Title: Effects of Parent-Implemented Video Self-Modeling on Conversational and Play Skills of Young Children With Developmental Delays
Brief Title: Home-Based Social Skills Intervention for Young Children With Developmental Delays
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNLV-2023-356
Record Dates: First submitted 2023-12-04; First posted 2023-12-28 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Development Delay; Social Skills; Parents
MeSH Terms: conditions — Learning Disabilities; Social Skills

STUDY DESIGN:
Intervention Model Description: The study will be a single subject design which will be replicated across multiple participants. The participants are pairs of one parent and one child for each session. The participants will be observed during the initial baseline phase before the intervention. The baseline phase will be used to compare the initial abilities before the intervention of the participants to their abilities after the intervention. After the baseline, the parent will participate in a parent training on how to use video modeling intervention with their child. Then the intervention phase begins. The parent and child will watch the video created to show new play skills for the child together and then have a play session. The parent will receive coaching before and after sessions.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Parent-Implemented Video Modeling (Experimental): Parent intervention teaches the skills to implement video modeling intervention for their young child with a developmental delay. Video modeling intervention teaches the young child new play and conversation skills.
  Interventions: Behavioral: Parent Training; Behavioral: Video Modeling

INTERVENTIONS:
Behavioral: Parent Training — Parent training will cover the topic of creating social skills, goal setting, creating a video model, how to implement the video model intervention, and the parent-child interaction procedures during play. Parents will learn the steps in the fidelity checklist and demonstrate the steps at 90% proficiency by the end of the training. Parent coaching will continue before and after child intervention sessions.
Behavioral: Video Modeling — The child will be recorded for a video model engaging in play at their home. The videos will be created with the parent and researcher in the home. A video using the same materials in the same location will be created depicting the child in a play scenario. The video will be two-to-three minutes in length. Each child will receive at least three sessions of intervention and no more than five sessions of intervention per week.

SUMMARY:
The goal of this clinical trial is to learn about how parent training can be used to teach a social skills intervention for their young child with developmental delays. Video modeling is a type of technology based intervention that teaches new skills using videos of someone acting out the behavior. The main questions it aims to answer are:

* How well do the parent training procedures teach parents all the steps for using video modeling as a social skills intervention?
* Do the children with developmental delays play and communicate more with their parents after the parent uses video modeling as a social skills intervention?

Parent participants will be asked to participate in 3 interviews 30 min to 1 hour each, 2 in-home sessions 1 ½ to 2 hours each, 30 min Zoom sessions 2-3 times per week for 2-5 months

Child participants will participate in 2 in-home sessions 1 ½ to 2 hours each and 30 min Zoom sessions 2-3 times per week for 2-5 months

The time commitment is in ideal conditions, but will be impacted by other participants and parent schedules. The family will be committing to approximately 2-5 hours per week for 2-5 months. Sessions may occur as few as 0 or as many as 5 times per week.

The hypothesis is that the parent training will teach parents all the steps to use video modeling intervention in their home with their young child with a disability. The second hypothesis is that the child with a disability will learn new social skills to play and communicate better in their home with their parent after watching the video models.

DETAILED DESCRIPTION:
Research Questions

1. What are the effects of video model training for parents on implementation fidelity of video self-modeling intervention for play actions and vocalizations for their young children with disabilities?
2. What are the effects of parent-implemented video self-modeling on play actions and vocalizations of young children with disabilities? Video self-modeling (VSM) is a type of video modeling that uses the person themselves acting out the behavior in the video. Hypothesis for question 1 is that the video model training provided to parents will increase their ability to implement steps of the intervention with fidelity. The hypothesis for question 2 is the parent-implemented video self-modeling intervention will increase the child's use of scripted and unscripted play actions and increase the child's use of scripted and unscripted verbalizations during play.

Methods

The design for the proposed study will be single subject multiple baseline across participants to answer the research questions 1 and 2. Replication across participants will allow for the verification of effects of the intervention. The study will consist of three phases: baseline, intervention, and maintenance. Baseline observes the behaviors before intervention begins. Intervention phase will teach the new behaviors for parent and child. Last maintenance measures the behaviors after they have been taught. Each participant will have pre assessments conducted before the baseline phase. The family home will be used as the setting for the study.

Procedures

Pre-assessment and Initial Home Visit

Before the baseline phase, the researcher will conduct the first of two in-home visits for the family. In the first home visit, the researcher will conduct pre-assessments to determine the social skills level and language development of the child. Pre-assessment session will include administering the Ages & Stages Questionnaires®, Third Edition (ASQ-3; Squires & Bricker, 2009) and Ages & Stages Questionnaires®: Social-Emotional, Second Edition (ASQ:SE-2; Squires et al., 2015), assessment of imitation skills, and ability to attend to a video. The ASQ-3 and the ASQ:SE-2 assess the developmental levels for young children between birth and five and half years old. The ASQ:SE-2 focuses on social and emotional development specifically. Each of the ASQ assessments take about 10-15 minutes to complete with parent report of child's current performance of tasks. The assessment to assess imitation skills will involve 20 trials of physical movements to imitate and 20 trials of verbalizations to imitate. The researcher will say, "do this" or "say this" followed by behavior as initial instructions for imitation. The child will need to imitate at least 10 physical movements and 10 verbalizations. The child will also be assessed on the ability to view a screen. The child will be given a preferred video based on parent report. The child needs to attend to the video for at least 5 minutes.

After pre-assessments are completed to ensure the child meets the criterion of participation, a preference assessment will be completed in the home to choose materials. The preference assessment will be naturalistic free operant observation in which the child will be given free access to toys in their home for 5 minutes (Cooper, 2020). The researcher will record the amount of time the child plays with each item in the 5 minutes. The researcher and parent will decide the best materials to use for the child based on parent report and preference assessment. Once materials are selected, the family will decide a location in the house for the play sessions to occur. The play sessions should occur in an area of the house where play typically occurs. The child should only have access to the chosen materials during the play sessions. The researcher will give parents instructions about how to conduct the play sessions with baseline procedures. The parent will practice a 10-minute session with researcher feedback to ensure the parent is not prompting the child during play sessions. The initial in-home session will conclude with a review of the procedures for baseline, schedule the next appointment, and ask parents if they have any questions.

Baseline

During the baseline phase, data will be collected via virtual sessions using a webcam, microphone, and video conferencing software, such as Zoom. The family will arrange the play area with the predetermined materials, so the child can access only the selected materials. The parent will set up a computer to record video and audio in a live stream session with the researcher. The device should be set up in a manner that allows the camera a clear view of the play area and the microphone close enough to hear both participants. Before the play session, the parent and researcher will have an informal interview to build rapport and collect field notes. The researcher will also address any questions and/or concerns of the parent during the initial conversation before play. The researcher will conduct a short coaching session to review the procedures. At the beginning of the 10-minute play session, the parent will instruct the child, "Let's play." The parent and the child will conduct a play session for ten minutes. The parent will be instructed to not prompt the child when playing, but the parent could prompt the child to stay in the play area. Data will be collected for five minutes of the play session at least two minutes after the session starts. Frequency data will be used to assess the number of actions and number of vocalizations during play. The researcher will be a nonparticipant observer during the 10-minute play session. After the baseline play session ends, another informal conversation with the parent and researcher will take place. The researcher will thank the family for their time, schedule the next appointment, and give positive feedback to the parent. The researcher will ask the parent if they have any questions. Field notes will be collected during each session to measure social validity.

Parent Training In-Home

Initial parent training will occur between the baseline and intervention phases. The researcher will conduct the parent training as the second in-home visit. Initial training has three goals: (1) choose play sequences and vocalizations, (2) collect footage for VSM with scripted actions and vocalizations, and (3) implement VSM intervention with >90% implementation fidelity. The parent training will consist of creating a social goal and scenario for the child based on the parent input and child preferences, creating the VSM video model, and practicing the fidelity checklist.

First, the researcher and parent will create the goal and scenario that will be appropriate for developmental levels and age-appropriate play and conversational skills. The researcher and parent will work together to create verbalizations and scripted play actions to interact with selected materials and the parent.

Once the script is written, VSM will be shot using the child as the model. A device with the capability to record video and audio with video editing software will be used to create the VSM videos, such as a tablet. Examples of video editing software include Google photos and iMovie. The parent and researcher will prompt the child to imitate the verbalizations and actions chosen by the parent and researcher. Each of the actions will be video recorded and then edited together a two-to-three-minute video. The same materials will be used from baseline with scripted play actions and vocalizations.

The third objective, the researcher and parent will review the fidelity checklist. The parent will learn how to respond to the child in a way that naturally reinforces social interaction instead of structured reinforcement schedules or prompting. The parent will practice implementing the fidelity checklist with the researcher to achieve 90% during the training process. The parent and child will view a preferred video to practice the video modeling procedures, then practice transitioning procedures to the play area. The play session will be 10-minutes, similar to the baseline sessions, but the parent will have more skills to demonstrate. The researcher will give corrective prompting and positive feedback during the session to achieve 90% or more during the initial parent training. The parent training will take approximately one hour in the family home. After the training, intervention phase will be scheduled, parent will be asked if they have any questions, and informal conversation. Field notes will be created and video recording of initial parent training will be data collected for fidelity and social validity.

Intervention

During the intervention phase, sessions will be conducted similarly to the baseline phase using virtual sessions. Video and audio equipment should be set up to view the parent and child during video viewing and the play session. Before VSM intervention and the play session, the researcher will have a conversation with the parent to review the fidelity checklist and ask the parent if they have any questions.

Once the intervention and play session begin, the researcher will then become an observer. The parent will have the child in a predetermined location to watch the video. The location chosen should be free of distraction and comfortable for the child. The parent will ensure the child is in the predesignated area for the viewing of the video. The parent will show the video clip to their child twice. The parent will say, "Let's watch a video." The parent will not say anything else until the end of the video viewing session. The only exception would be to redirect the child to attend to the video. The parent will end the video viewing with praise (e.g. "Great job, watching the video"). Then a transition between the video viewing area and the play area will occur.

The play session will begin with the parent saying, "Let's play." The parent will implement the fidelity checklist during the video viewing and the play session. The parent will be instructed to provide no prompting. The only exception will be to prompt the child to stay in the play area. The parent will use natural reinforcement techniques to engage the child while playing. The parent will respond to the child within 3 seconds of initiation, comment, or play action. The parent will demonstrate skills during play. Based on fidelity checklist the researcher will determine the percentage of steps the parent followed throughout the session. The child and parent will play for 10 minutes. Data on the four child outcomes will be collected each session along with dependent variables for parent fidelity.

Once the parent implements the intervention at 80% accuracy or higher for three consecutive sessions, the maintenance phase will begin. The intervention phase may also end if the child has achieved 80% of scripted play actions and scripted vocalizations for 3 sessions. During the intervention phase, the parent will participate in the second of three interviews to collect data about their perspectives about the intervention to assess social validity of the program.

Maintenance

Once the intervention phase ends, the parent and child dyad will move into maintenance phase. Follow-up will occur 2 weeks and 4 weeks after the end of the intervention. Procedures for the follow-up phase will match the baseline procedures. Data will be collected for the parent's fidelity for implementing the play session using natural reinforcements and modeling. The child will have data collected for the four dependent variables: scripted and unscripted play action and vocalizations. In addition, the parents will participate in the last interview via video call to collect data on the social validity of the intervention process.

ELIGIBILITY:
Inclusion Criteria

Parent

* English speaking
* Must to participate in in-home parent training, willing to participate in video interviews, willing to participate in video recorded play sessions
* Only one parent in the home will participate
* At least 18 years old and able to consent to participate in study

Child

* between the ages 3 and 5.5
* have a developmental delay as defined by Individuals with Disability Education Act
* demonstrate a need for social skills intervention with ASQ:SE-2 scoring below cutoff or in the monitoring zone.
* shows the ability to use 1 to 2-word phrases
* imitates 10 actions and 10 words
* attends to a video for 3 minutes

Exclusion criteria

* English is not a primary language spoken at home
* the home is unsafe (Defined as violence witnessed in the home, drug or alcohol use while researcher is in the home, and non-service animals in the intervention area.)
* the child does not display minimum levels of language (e.g., 1 to 2 word phrases), imitation (e.g., 10 gestures 10 words) and/or attention (e.g., 3 minutes attending to a screen)
* the child does not show social skills delays ASQ:SE-2 scoring above the cutoff.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Parent: Implementation Fidelity | Implementation fidelity data will be collected for 5 minutes during a session, 2-3 times per week for 2 to 5 months in ideal conditions. To adjust for parent schedules and commitments, as few as 0 to as many as 5 sessions per week may be conducted.
  For parent behavior, the dependent variable that will be measured will be the percentage of implementation fidelity based on the procedural checklist for the intervention. The parent will implement the intervention and conduct play sessions. The checklist includes how the parents will set up the physical environment for viewing the video and for play sessions. The parent will follow a guide for parent-child interaction to control for variables like prompting.
Child: Scripted Play Actions | Scripted play action data will be collected for 5 minutes during a session, 2-3 times per week for 2 to 5 months in ideal conditions. To adjust for parent schedules and commitments, as few as 0 to as many as 5 sessions per week may be conducted.
  For child behavior, frequency of scripted play actions will be measured. Scripted play actions defined as motor movements with or without materials in the play area that make sense within the context of play and portrayed in the video model. Frequency data will be collected for 5 minutes. Stereotyped movements will not be recorded in the frequency.
Child: Unscripted Play Actions | Unscripted play action data will be collected for 5 minutes during a session, 2-3 times per week for 2 to 5 months in ideal conditions. To adjust for parent schedules and commitments, as few as 0 to as many as 5 sessions per week may be conducted.
  For child behavior, frequency of scripted play actions will be measured. For child behavior, frequency of unscripted play actions will be measured. Unscripted play actions defined as motor movements with or without materials in the play area that make sense within the context of play and are not portrayed in the video model. Frequency data will be collected for 5 minutes. Stereotyped movements will not be recorded in the frequency.
Child: Scripted Vocalizations | Scripted vocalization data will be collected for 5 minutes during a session, 2-3 times per week for 2 to 5 months in ideal conditions. To adjust for parent schedules and commitments, as few as 0 to as many as 5 sessions per week may be conducted.
  For child behavior, frequency of scripted vocalizations will be measured. Scripted vocalizations defined as words, short phrases, and play sounds (e.g. "vroom", "whoosh") that make sense in the context of play and portrayed in the video model. Frequency data will be collected for 5 minutes. Repetitive sounds or words will only be recorded once.
Child: Unscripted Vocalizations | Unscripted vocalization data will be collected for 5 minutes during a session, 2-3 times per week for 2 to 5 months in ideal conditions. To adjust for parent schedules and commitments, as few as 0 to as many as 5 sessions per week may be conducted.
  For child behavior, frequency of unscripted vocalizations will be measured. Unscripted vocalizations defined as words, short phrases, and play sounds (e.g. "vroom", "whoosh") that make sense in the context of play and are not portrayed in the video model. Frequency data will be collected for 5 minutes. Repetitive sounds or words will only be recorded once.

CONTACTS AND LOCATIONS:
Overall Officials: Alain Bengochea, PhD, Principal Investigator — University of Nevada, Las Vegas
Locations (1):
- University of Nevada, Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cooper, J. 0., Heron, T. E., & Heward, W. L. (2020). Applied behavior analysis (3rd edition). Pearson: Hoboken, NJ.
- [Background] Squires, J. & Bricker, D. (2009). Ages & Stages Questionnaires®, (3rd ed., ASQ®-3): A parent-completed child monitoring system. Paul H. Brookes Publishing Co., Inc.
- [Background] Squires, J., Bricker, D., & Twombly, E. (2015) Ages & Stages Questionnaires®: Social-emotional (2nd ed., ASQ®:SE-2): A parent-completed child monitoring system for social-emotional behaviors. Paul H. Brookes Publishing Co., Inc.